CLINICAL TRIAL: NCT01656070
Title: Vitamin D Status and T Cell Phenotype in HIV-infected Youth Supplemented With Cholecalciferol: a Randomized Clinical Trial.
Brief Title: Vitamin D Supplementation in HIV-infected Youth
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Milan (Other)
Responsible Party: Principal Investigator, Gian Vincenzo Zuccotti, Gian Vincenzo Zuccotti, Associate Professor of Pediatrics, Chief of Department of Pediatrics at L. Sacco Hospital, University of Milan
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HLS02/2011-1.0-09-11-2010; 2011-000593-54 (EudraCT Number)
Record Dates: First submitted 2012-07-31; First posted 2012-08-02 (Estimated); Last update posted 2012-08-02 (Estimated); Status verified 2012-08

CONDITIONS: HIV Disease; Vitamin D Deficiency; Hypovitaminosis D; Hyperparathyroidism
Keywords: HIV; children; adolescents; Vitamin D; immunity; T cell phenotype
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Vitamin D Deficiency; Hyperparathyroidism | interventions — Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Vitamin D (Experimental): oral cholecalciferol 1000000 UI (vitamin D3).
  At 0, 3, 6 and 9 months, the vitamin D group received orally 100000 IU of cholecalciferol suspended in 2 mL of olive oil in sealed plastic syringes labeled with the unique identification numbers.
  Interventions: Drug: oral cholecalciferol 1000000 UI (vitamin D3)
- placebo (Placebo Comparator): placebo
  At 0, 3, 6 and 9 months, the placebo group received 2 mL of olive oil, in sealed plastic syringes labeled with the unique identification numbers.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: oral cholecalciferol 1000000 UI (vitamin D3)
  Other Names: DIBASE - ABIOGEN PHARMA Spa
  Arms: Vitamin D
Drug: Placebo
  Arms: placebo

SUMMARY:
Along with its effects on bone metabolism, vitamin D is an important modulator of the immune system. Experimental studies have shown that the active metabolite of vitamin D [1,25(OH)2D] is able to skew the T cell compartment into a more anti-inflammatory state, with inhibition of Th1 and Th17 cells and promotion of Th2 and T regulatory subsets.

In the context of HIV infection, in which Th1 subpopulations are devoted to inhibit viral replication, any alteration of the Th1/Th2 balance would be of concern.

The aim of this Randomized Controlled Trial is to test wether oral supplementation with cholecalciferol could be able: 1) to improve vitamin D status and, 2) to play an immunomodulatory role, in vertically HIV-infected children and young adults with hypovitaminosis D.

DETAILED DESCRIPTION:
There is increasing evidence that hypovitaminosis D is common in the general population.

Low dietary intake of vitamin D and reduced exposure to sunlight are probably the major risk factors. A high prevalence of hypovitaminosis D has been described in HIV-infected adults, and children. HIV infection itself and antiretroviral (ARV) treatment may be responsible for alteration of vitamin D metabolism. For instance, studies have shown a significant decrease in serum 25-hydroxyvitamin-D [25(OH)D] concentration in adults receiving non-nucleoside reverse transcriptase inhibitors (NNRTIs). Whatever the cause(s) of hypovitaminosis D, because of the importance of vitamin D in bone health, randomized controlled trials (RCT) have been performed to test whether vitamin D supplementation can improve vitamin D status and bone mineral metabolism in HIV-infected children and adolescents.

Along with its effects on bone metabolism, vitamin D is an important modulator of the immune system. The vitamin D receptor (VDR) is found in high concentrations in activated T lymphocytes, in small amounts in monocyte/macrophage cells while B lymphocytes do not contain detectable amounts of VDR.

Experimental studies have shown that the active di-hydroxylated metabolite of vitamin D [1,25(OH)2D] is able to skew the T cell compartment into a more anti-inflammatory state, with inhibition of Th1 and Th17 cells and promotion of Th2 and T regulatory (Treg) subsets.

In the context of HIV infection, in which Th1 subpopulations are devoted to inhibit viral replication, 16 any alteration of the Th1/Th2 balance would be of concern.

Although all the biological effects of vitamin D are mediated by the 1,25(OH)2D, it is the 25(OH)D to be routinely quantified because of its longer half-life.17 However, HIV-infected subjects may have a defective 1α-hydroxylation of 25(OH)D. Thus, it is important to evaluate the effects of vitamin D supplementation both in terms of 25(OH)D and 1,25(OH)2D responses.

This repeated-measures parallel-group RCT is aimed to test wether a 12-month oral supplementation with cholecalciferol (vitamin D3) is able: 1) to increase serum 25(OH)D and 1,25(OH)2D levels and, 2) to affect T-cell phenotype in vertically HIV-infected children and young adults with hypovitaminosis D and stable HIV-disease.

Main outcome: to determine the frequency of hypovitaminosis D at 12-month of follow-up among subjects supplemented with oral cholecalciferol versus subjects receiving placebo.

Secondary outcome: to investigate correlations - if any - between serum vitamin D concentration and markers of immune activation (i.e. Th1-, Th2-, Th17- and Treg-lymphocytes count, T-lymphocyte VDR expression)

ELIGIBILITY:
Inclusion Criteria:

* Vertically acquired HIV infection
* age < 30 years
* serum 25(OH)D concentration < 30 ng/mL
* signed written informed consent

Exclusion Criteria:

* hyperparathyroidism, as detected by an intact serum parathyroid hormone (PTH) ≥ 65 pg/mL
* Black ethnic group
* any supplementation with vitamin D in the previous 12 months
* use of any treatment known to alter vitamin D status in the previous 6 months (excluding ARV)
* any concomitant severe illness.

Max Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 50 (Actual)
Dates: Start 2011-04; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
frequency of Hypovitaminosis D [serum 25(OH)D < 30 ng/mL] in the Vitamin D receiving group vs placebo group | 12 months
  Vertically HIV-infected patients aged <30 years and with serum 25(OH)D < 30 ng/mL were randomized into the vitamin D or placebo group. At baseline (0 months), 3, 6 and 9 months, the intervention group received orally 100000 IU of cholecalciferol. Serum 25(OH)D, 1,25(OH)2D, PTH and CD4+ T cells were assessed 3 months before baseline, at 0, 3, 6, 9 and 12 months, while Th1-, Th2-, Th17- and Treg-subsets and T-lymphocyte vitamin D receptor at 0, 3 and 12 months

SECONDARY OUTCOMES:
Effect of oral cholecalciferol supplementation on T cell phenotype in vertically HIV-infected youth with stable HIV diseases | 12 months
  Vertically HIV-infected patients aged <30 years and with serum 25(OH)D < 30 ng/mL were randomized into the vitamin D or placebo group. At baseline (0 months), 3, 6 and 9 months, the intervention group received orally 100000 IU of cholecalciferol. CD4+ T-cells were assessed 3 months before enrollment (-3 months), at baseline (0 months) and at each visit thereafter (3, 6, 9 and 12 months). T-lymphocyte VDR expression and Th1-, Th2-, Th17- and Treg-lymphocytes were measured at 0, 3 and 12 months.

CONTACTS AND LOCATIONS:
Overall Officials: Gian Vincenzo Zuccotti, Professor, Principal Investigator — Department of Paediatrics, L. Sacco Hospital, University of Milan, Milan, Italy
Locations (1):
- Department of Paediatrics - L. Sacco Hospital, Milan, Italy

REFERENCES:
- [Background] Zadshir A, Tareen N, Pan D, Norris K, Martins D. The prevalence of hypovitaminosis D among US adults: data from the NHANES III. Ethn Dis. 2005 Autumn;15(4 Suppl 5):S5-97-101. PMID 16315387
- [Background] Bischoff-Ferrari HA. "Vitamin D - why does it matter?" - defining vitamin D deficiency and its prevalence. Scand J Clin Lab Invest Suppl. 2012;243:3-6. doi: 10.3109/00365513.2012.681938. PMID 22536756
- [Background] Kuehn EW, Anders HJ, Bogner JR, Obermaier J, Goebel FD, Schlondorff D. Hypocalcaemia in HIV infection and AIDS. J Intern Med. 1999 Jan;245(1):69-73. doi: 10.1046/j.1365-2796.1999.00407.x. PMID 10095819
- [Background] Rodriguez M, Daniels B, Gunawardene S, Robbins GK. High frequency of vitamin D deficiency in ambulatory HIV-Positive patients. AIDS Res Hum Retroviruses. 2009 Jan;25(1):9-14. doi: 10.1089/aid.2008.0183. PMID 19108690
- [Background] Stephensen CB, Marquis GS, Kruzich LA, Douglas SD, Aldrovandi GM, Wilson CM. Vitamin D status in adolescents and young adults with HIV infection. Am J Clin Nutr. 2006 May;83(5):1135-41. doi: 10.1093/ajcn/83.5.1135. PMID 16685057
- [Background] Rutstein R, Downes A, Zemel B, Schall J, Stallings V. Vitamin D status in children and young adults with perinatally acquired HIV infection. Clin Nutr. 2011 Oct;30(5):624-8. doi: 10.1016/j.clnu.2011.02.005. Epub 2011 Jun 8. PMID 21641097
- [Background] Van Den Bout-Van Den Beukel CJ, Fievez L, Michels M, Sweep FC, Hermus AR, Bosch ME, Burger DM, Bravenboer B, Koopmans PP, Van Der Ven AJ. Vitamin D deficiency among HIV type 1-infected individuals in the Netherlands: effects of antiretroviral therapy. AIDS Res Hum Retroviruses. 2008 Nov;24(11):1375-82. doi: 10.1089/aid.2008.0058. PMID 18928396
- [Background] Mueller NJ, Fux CA, Ledergerber B, Elzi L, Schmid P, Dang T, Magenta L, Calmy A, Vergopoulos A, Bischoff-Ferrari HA; Swiss HIV Cohort Study. High prevalence of severe vitamin D deficiency in combined antiretroviral therapy-naive and successfully treated Swiss HIV patients. AIDS. 2010 May 15;24(8):1127-34. doi: 10.1097/QAD.0b013e328337b161. PMID 20168200
- [Background] Allavena C, Delpierre C, Cuzin L, Rey D, Viget N, Bernard J, Guillot P, Duvivier C, Billaud E, Raffi F. High frequency of vitamin D deficiency in HIV-infected patients: effects of HIV-related factors and antiretroviral drugs. J Antimicrob Chemother. 2012 Sep;67(9):2222-30. doi: 10.1093/jac/dks176. Epub 2012 May 15. PMID 22589455
- [Background] Conesa-Botella A, Florence E, Lynen L, Colebunders R, Menten J, Moreno-Reyes R. Decrease of vitamin D concentration in patients with HIV infection on a non nucleoside reverse transcriptase inhibitor-containing regimen. AIDS Res Ther. 2010 Nov 23;7:40. doi: 10.1186/1742-6405-7-40. PMID 21092280
- [Background] Arpadi SM, McMahon D, Abrams EJ, Bamji M, Purswani M, Engelson ES, Horlick M, Shane E. Effect of bimonthly supplementation with oral cholecalciferol on serum 25-hydroxyvitamin D concentrations in HIV-infected children and adolescents. Pediatrics. 2009 Jan;123(1):e121-6. doi: 10.1542/peds.2008-0176. PMID 19117833
- [Background] Arpadi SM, McMahon DJ, Abrams EJ, Bamji M, Purswani M, Engelson ES, Horlick M, Shane E. Effect of supplementation with cholecalciferol and calcium on 2-y bone mass accrual in HIV-infected children and adolescents: a randomized clinical trial. Am J Clin Nutr. 2012 Mar;95(3):678-85. doi: 10.3945/ajcn.111.024786. Epub 2012 Jan 18. PMID 22258265
- [Background] Veldman CM, Cantorna MT, DeLuca HF. Expression of 1,25-dihydroxyvitamin D(3) receptor in the immune system. Arch Biochem Biophys. 2000 Feb 15;374(2):334-8. doi: 10.1006/abbi.1999.1605. PMID 10666315
- [Background] Sloka S, Silva C, Wang J, Yong VW. Predominance of Th2 polarization by vitamin D through a STAT6-dependent mechanism. J Neuroinflammation. 2011 May 24;8:56. doi: 10.1186/1742-2094-8-56. PMID 21605467
- [Background] Baeke F, Takiishi T, Korf H, Gysemans C, Mathieu C. Vitamin D: modulator of the immune system. Curr Opin Pharmacol. 2010 Aug;10(4):482-96. doi: 10.1016/j.coph.2010.04.001. Epub 2010 Apr 27. PMID 20427238
- [Background] Klein SA, Dobmeyer JM, Dobmeyer TS, Pape M, Ottmann OG, Helm EB, Hoelzer D, Rossol R. Demonstration of the Th1 to Th2 cytokine shift during the course of HIV-1 infection using cytoplasmic cytokine detection on single cell level by flow cytometry. AIDS. 1997 Jul 15;11(9):1111-8. doi: 10.1097/00002030-199709000-00005. PMID 9233457
- [Background] Holick MF, Binkley NC, Bischoff-Ferrari HA, Gordon CM, Hanley DA, Heaney RP, Murad MH, Weaver CM; Endocrine Society. Evaluation, treatment, and prevention of vitamin D deficiency: an Endocrine Society clinical practice guideline. J Clin Endocrinol Metab. 2011 Jul;96(7):1911-30. doi: 10.1210/jc.2011-0385. Epub 2011 Jun 6. PMID 21646368
- [Background] Haug CJ, Aukrust P, Haug E, Morkrid L, Muller F, Froland SS. Severe deficiency of 1,25-dihydroxyvitamin D3 in human immunodeficiency virus infection: association with immunological hyperactivity and only minor changes in calcium homeostasis. J Clin Endocrinol Metab. 1998 Nov;83(11):3832-8. doi: 10.1210/jcem.83.11.5270. PMID 9814454
- [Background] Ryan P. Random allocation of treatments in blocks. Stata Journal;8:594, 2008
- [Background] Rabe-Hesketh S, Skrondal A. Multilevel and longitudinal modeling using Stata. Volume 1: Continuous responses. College Station, TX: Stata Press; 2012.
- [Background] Jacobson DL, Spiegelman D, Duggan C, Weinberg GA, Bechard L, Furuta L, Nicchitta J, Gorbach SL, Miller TL. Predictors of bone mineral density in human immunodeficiency virus-1 infected children. J Pediatr Gastroenterol Nutr. 2005 Sep;41(3):339-46. doi: 10.1097/01.mpg.0000174468.75219.30. PMID 16131991
- [Background] Signorello LB, Shi J, Cai Q, Zheng W, Williams SM, Long J, Cohen SS, Li G, Hollis BW, Smith JR, Blot WJ. Common variation in vitamin D pathway genes predicts circulating 25-hydroxyvitamin D Levels among African Americans. PLoS One. 2011;6(12):e28623. doi: 10.1371/journal.pone.0028623. Epub 2011 Dec 21. PMID 22205958
- [Background] Haug C, Muller F, Aukrust P, Froland SS. Subnormal serum concentration of 1,25-vitamin D in human immunodeficiency virus infection: correlation with degree of immune deficiency and survival. J Infect Dis. 1994 Apr;169(4):889-93. doi: 10.1093/infdis/169.4.889. PMID 7907645
- [Background] Teichmann J, Stephan E, Lange U, Discher T, Friese G, Lohmeyer J, Stracke H, Bretzel RG. Osteopenia in HIV-infected women prior to highly active antiretroviral therapy. J Infect. 2003 May;46(4):221-7. doi: 10.1053/jinf.2002.1109. PMID 12799147
- [Background] Kakalia S, Sochett EB, Stephens D, Assor E, Read SE, Bitnun A. Vitamin D supplementation and CD4 count in children infected with human immunodeficiency virus. J Pediatr. 2011 Dec;159(6):951-7. doi: 10.1016/j.jpeds.2011.06.010. Epub 2011 Aug 4. PMID 21820130
- [Background] Boonstra A, Barrat FJ, Crain C, Heath VL, Savelkoul HF, O'Garra A. 1alpha,25-Dihydroxyvitamin d3 has a direct effect on naive CD4(+) T cells to enhance the development of Th2 cells. J Immunol. 2001 Nov 1;167(9):4974-80. doi: 10.4049/jimmunol.167.9.4974. PMID 11673504
- [Background] Fazekas de St Groth B, Landay AL. Regulatory T cells in HIV infection: pathogenic or protective participants in the immune response? AIDS. 2008 Mar 30;22(6):671-83. doi: 10.1097/QAD.0b013e3282f466da. No abstract available. PMID 18356596
- [Background] Aandahl EM, Michaelsson J, Moretto WJ, Hecht FM, Nixon DF. Human CD4+ CD25+ regulatory T cells control T-cell responses to human immunodeficiency virus and cytomegalovirus antigens. J Virol. 2004 Mar;78(5):2454-9. doi: 10.1128/jvi.78.5.2454-2459.2004. PMID 14963140
- [Background] Sousa AE, Carneiro J, Meier-Schellersheim M, Grossman Z, Victorino RM. CD4 T cell depletion is linked directly to immune activation in the pathogenesis of HIV-1 and HIV-2 but only indirectly to the viral load. J Immunol. 2002 Sep 15;169(6):3400-6. doi: 10.4049/jimmunol.169.6.3400. PMID 12218162
- [Background] Bang U, Kolte L, Hitz M, Dam Nielsen S, Schierbeck LL, Andersen O, Haugaard SB, Mathiesen L, Benfield T, Jensen JE. Correlation of increases in 1,25-dihydroxyvitamin D during vitamin D therapy with activation of CD4+ T lymphocytes in HIV-1-infected males. HIV Clin Trials. 2012 May-Jun;13(3):162-70. doi: 10.1310/hct1303-162. PMID 22592096
- [Background] D'Ambrosio D, Cippitelli M, Cocciolo MG, Mazzeo D, Di Lucia P, Lang R, Sinigaglia F, Panina-Bordignon P. Inhibition of IL-12 production by 1,25-dihydroxyvitamin D3. Involvement of NF-kappaB downregulation in transcriptional repression of the p40 gene. J Clin Invest. 1998 Jan 1;101(1):252-62. doi: 10.1172/JCI1050. PMID 9421488
- [Background] Shearer GM, Clerici M. Cytokine profiles in HIV type 1 disease and protection. AIDS Res Hum Retroviruses. 1998 Jun;14 Suppl 2:S149-52. No abstract available. PMID 9672232
- [Background] Clerici M, Seminari E, Maggiolo F, Pan A, Migliorino M, Trabattoni D, Castelli F, Suter F, Fusi ML, Minoli L, Carosi G, Maserati R; Master Group. Early and late effects of highly active antiretroviral therapy: a 2 year follow-up of antiviral-treated and antiviral-naive chronically HIV-infected patients. AIDS. 2002 Sep 6;16(13):1767-73. doi: 10.1097/00002030-200209060-00009. PMID 12218388